CLINICAL TRIAL: NCT00001620
Title: Screening Protocol for Subjects Being Evaluated for National Heart, Lung and Blood Institute (NHLBI) Protocols
Brief Title: Screening for Hematology Branch Protocols
Status: Enrolling by invitation | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970041; 97-H-0041
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-21

CONDITIONS: Hematologic Disease and Disorders; Donors; Healthy Volunteer
Keywords: Thrombocytopenia; Anemia; Neutropenia; Dysplasia; Hematopoiesis; Cytopenia; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Diseases; Disease; Thrombocytopenia; Anemia; Neutropenia; Cytopenia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects undergoing screening: Adults and children being screened for an active NHLBI protocol

SUMMARY:
This study allows the evaluation of subjects in order to determine their ability to safely participate in other active research studies.

After subjects complete the screening process, they will be offered the opportunity to participate in an active research study, or if no appropriate studies are available information and recommendations will be provided for other treatment options.

DETAILED DESCRIPTION:
This protocol is designed for screening of subjects before a decision can be made as to their eligibility for one of the active National Heart, Lung, and Blood Institute (NHLBI) research protocols. Its purpose is to allow detailed investigation into the hematologic or oncologic problems of these subjects, and the status of other organ systems that would determine their ability to safely tolerate specific aspects of active research protocols. It allows investigation as to whether a donor is HLA matched, fit to receive G-CSF, and fit to undergo apheresis and therefore eligible to participate as a donor on a bone marrow transplant protocol. It also allows the investigation as to whether subjects are eligible for participation as normal volunteer based on protocol eligibility criteria that requires generally good health status by history or physical exam findings, or laboratory assessments. After completion of this screening process, the subject will either be offered a chance to participate in an active research protocol, or if no appropriate protocol is identified, subjects with hematologic or oncologic disease will have recommendations for other treatment options relayed to the primary or referring physician.

Primary objective is to determine subject eligibility for participation on NHLBI protocols.

Primary endpoint is the results of clinical, imaging and laboratory assessments.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be entered on this protocol at the time of their first visit to the NIH Clinical Center outpatient clinic or inpatient service if:

The subject carries the diagnosis of a disorder for which the NHLBI has an active research protocol, and based on information received from an outside physician, he/she appears to meet at least preliminary eligibility criteria for that protocol.

OR

The subject is a donor for a subject for which the NHLBI has an active stem cell transplant protocol and based on information received from an outside physician, he/she appears to meet preliminary eligibility as a donor.

OR

The subject is a normal volunteer for which the NHLBI has an active study recruiting healthy normal volunteers and he/she appears to meet preliminary eligibility as a normal volunteer.

Age greater than or equal to 2 and Weight greater than 12 kg. (Healthy Volunteer age greater than or equal to 8)

The subject, the subject s guardian (if the subject is a minor), or the subject s legally authorized representative (LAR) is capable of informed consent, and willing to sign the consent form after initial counseling by clinical staff. Separate consent forms for all interventional or surgical procedures will be obtained after explanation of the specific procedure.

EXCLUSION CRITERIA:

All subjects not fulfilling the inclusion criteria will be considered ineligible.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects referred for active National Heart, Lung, and Blood Institute (NHLBI) research protocols, donors and healthy volunteers@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1996-12-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the results of clinical, imaging and laboratory assessments. | ongoing
  Results of clinical, imaging and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balakrishna J, Basumallik N, Matulonis R, Scott D, Salem D, Jasper G, Wiestner A, Stetler-Stevenson M, Marti G, Sun C, Yuan CM. Intensity of antigen expression reflects IGHV mutational status and Dohner-defined prognostic categories in chronic lymphocytic leukemia, monoclonal B-cell lymphocytosis, and small lymphocytic lymphoma. Leuk Lymphoma. 2021 Aug;62(8):1828-1839. doi: 10.1080/10428194.2021.1894641. Epub 2021 Mar 18. PMID 33734005
- [Derived] Wu Z, Gao S, Diamond C, Kajigaya S, Chen J, Shi R, Palmer C, Hsu AP, Calvo KR, Hickstein DD, Holland SM, Young NS. Sequencing of RNA in single cells reveals a distinct transcriptome signature of hematopoiesis in GATA2 deficiency. Blood Adv. 2020 Jun 23;4(12):2656-2670. doi: 10.1182/bloodadvances.2019001352. PMID 32556286
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] Giudice V, Feng X, Lin Z, Hu W, Zhang F, Qiao W, Ibanez MDPF, Rios O, Young NS. Deep sequencing and flow cytometric characterization of expanded effector memory CD8+CD57+ T cells frequently reveals T-cell receptor Vbeta oligoclonality and CDR3 homology in acquired aplastic anemia. Haematologica. 2018 May;103(5):759-769. doi: 10.3324/haematol.2017.176701. Epub 2018 Feb 1. PMID 29419434
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-H-0041.html